CLINICAL TRIAL: NCT05587504
Title: Determination of Liquid Flavor and Nicotine Form Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HM20025474; U54DA036105 (NIH)
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Electronic Cigarettes
MeSH Terms: conditions — Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: Each participant will participate in 5 sessions. Sessions differ by the tobacco product used (see study arms). The sessions will be ordered by latin-square; however, session order is NOT expected to change any outcomes and order effects are not relevant to the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cigarette and/or e-Cigarette users (Experimental): Each participant will participate in 4 sessions. During each session, participants will first complete a 10-puff product use period with the ECIG assigned for that session, then a 30-minute ad lib product use period, and then a cigarette/e-cigarette challenge paradigm.
  Interventions: Other: E-cigarette with sweetness type 1 and pronation level 1; Other: E-cigarette with sweetness type 1 and pronation level 2; Other: E-cigarette with sweetness type 2 and pronation level 1; Other: E-cigarette with sweetness type 2 and pronation level 2

INTERVENTIONS:
Other: E-cigarette with sweetness type 1 and pronation level 1 — An "open system" ECIG (Kanger Sub Box Mini and/or a Kangertech Sub Box Mini tank connected to hardware and/or software to limit puff duration) set to 15 Watts, which will contain e-liquid that contains a predetermined mg/ml of nicotine and sweetness type 1 and protonation level 1.
Other: E-cigarette with sweetness type 1 and pronation level 2 — An "open system" ECIG (Kanger Sub Box Mini and/or a Kangertech Sub Box Mini tank connected to hardware and/or software to limit puff duration) set to 15 Watts, which will contain e-liquid that contains a predetermined mg/ml of nicotine and sweetness type 1 and protonation level 2.
Other: E-cigarette with sweetness type 2 and pronation level 1 — An "open system" ECIG (Kanger Sub Box Mini and/or a Kangertech Sub Box Mini tank connected to hardware and/or software to limit puff duration) set to 15 Watts, which will contain e-liquid that contains a predetermined mg/ml of nicotine and sweetness type 2 and protonation level 1.
Other: E-cigarette with sweetness type 2 and pronation level 2 — An "open system" ECIG (Kanger Sub Box Mini and/or a Kangertech Sub Box Mini tank connected to hardware and/or software to limit puff duration) set to 15 Watts, which will contain e-liquid that contains a predetermined mg/ml of nicotine and sweetness type 2 and protonation level 2.

SUMMARY:
The purpose of this research study is to find out how different types of electronic cigarette/vape e-liquids with differing sweetness and forms of nicotine affect blood nicotine levels, use behavior (how people puff), and how people feel.

DETAILED DESCRIPTION:
In this study, participants will be asked to do the following:

1. After an initial screening visit, visit the Center for the Study of Tobacco Products 4 more times for approximately 3-hour study visits.
2. Before each visit, abstain from all tobacco products (cigarettes, e-cigarettes/vapes, cigars, and hookah/waterpipe) for at least 12 hours.
3. Allow researcher to take blood pressure readings (with blood pressure cuff on their arm) monitor their heart rate (with a device that attaches to their finger), and allow a nurse to insert an IV catheter into their arm that will stay there for the entire session. This catheter will be used to draw blood periodically (less than 1 tablespoon per sample, 5 samples per visit).
4. During each session, participants will respond to several questionnaires to measure how they feel before and after they use an e-cigarette.
5. In each session, use an electronic cigarette provided by the study team at two separate times. After using the e-cigarette two times, participants will be offered the opportunity to use their own e-cigarette or cigarette.

ELIGIBILITY:
Inclusion Criteria:

* healthy (determined by self-report)
* between the ages of 18-65
* willing to provide informed consent
* use cigarettes, e-cigarettes, or both
* able to attend the lab and abstain from tobacco/nicotine as required and must agree to use designated products according to study protocol

Exclusion Criteria:

* women if they are breast-feeding or test positive for pregnancy (by urinalysis) at screening
* existence of any condition contraindicated for this study protocol as determined by study leadership

Some study details about the eligibility criteria are purposely omitted at this time to preserve scientific integrity. Full details will be posted at the conclusion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Change in plasma nicotine concentration | Baseline (approx 90 min after session start) to after final product usage (up to 165 min)
  Blood will be taken multiple times in each session to examine changes in plasma nicotine concentration from baseline to after various e-cigarette or cigarette usage.
Puff volume | Through the final product use (up to 165 min)
  The volume of each puff, in ml, averaged over each product use bout.
Puff duration | Through the final product use (up to 165 min)
  The duration of each puff, in ml, averaged over each product use bout.
Challenge paradigm latency | at the end of the challenge paradigm, approx. 165 min
  The cigarette or own brand e-cigarette challenge paradigm involves giving participants a five minute period to use their own brand cigarette or e-cigarette. Researchers measure the time it takes for the participant to pick up the product.
Challenge paradigm puffs | at the end of the challenge paradigm, approx. 165 min
  The cigarette or own brand e-cigarette challenge paradigm involves giving participants a five minute period to use their own brand cigarette or e-cigarette. Researchers measure the number of puffs the participant takes.

OTHER OUTCOMES:
Change in Direct Effects of Product use Questionnaires | Baseline (approx 90 min after session start) to after final product usage (up to 185 min)
  Surveys will be completed multiple times in each session to examine changes from baseline to after specific e-cigarette or cigarette usage.
  This scale is used to assess how product use makes participants feel and consists of 10 questions each for e-cigarettes and cigarettes that are scored 0 - 100. There are no sub-scales. Items are analyzed separately.
Change in Hughes-Hatsukami Questionnaire | Baseline (approx 90 min after session start) to after final product usage (up to 185 min)
  Surveys will be completed multiple times in each session to examine changes from baseline to after specific e-cigarette or cigarette usage.
  This scale will be used to assess the extent to which product use reduces tobacco abstinence symptoms, and consists of 11 items scored 0-100, with lower scores indicating less severe symptoms. There are no sub-scales. Items are analyzed separately.
Change in General Labeled Magnitude Scale | Baseline (approx 90 min after session start) to after final product usage (up to 185 min)
  Surveys will be completed multiple times in each session to examine changes from baseline to after specific e-cigarette or cigarette usage.
  This scale measures the flavor sensation, harshness, and throat hit (in three questions that correspond to those constructs) of the e-cigarette used in each session. The scale ranges from 0 - 100, with 0 being no sensation and 100 being the strongest imaginable sensation of any kind. Each item is scored and analyzed separately (there are no sub-scales).
Change in Labeled Hedonic Scale | Baseline (approx 90 min after session start) to after final product usage (up to 185 min)
  Surveys will be completed multiple times in each session to examine changes from baseline to after specific e-cigarette or cigarette usage.
  This measure is related to perceptions of electronic cigarette effects (4 questions, each scored from 0 - 100).

CONTACTS AND LOCATIONS:
Overall Officials: Alison Breland, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT05587504/ICF_000.pdf